CLINICAL TRIAL: NCT03043417
Title: Exploring Stigma, Discrimination, and Recovery-based Perspectives Toward Mental Illness and Substance Use Problems
Brief Title: Stigma Intervention Among Primary Health Workers in Toronto
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Akwatu Khenti, Director, Global Health, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 0512014
Record Dates: First submitted 2016-12-14; First posted 2017-02-06 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Mental Health Disorder; Substance Use
Keywords: Stigma; Primary Health Care; Recovery
MeSH Terms: conditions — Mental Disorders; Substance-Related Disorders; Social Stigma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CHC's given the intervention (Experimental): Three CHC sites where all staff receive all components of the intervention. Training, Media, Art workshops, and a Policy analysis as well as survey completion.
  Interventions: Behavioral: CHC's given the intervention
- CHC's with NO intervention (No Intervention): Three CHC sites where all staff and a selection of clients complete surveys but receive no intervention.

INTERVENTIONS:
Behavioral: CHC's given the intervention — CHC's NOT given the intervention
  Arms: CHC's given the intervention

SUMMARY:
This project is measuring the effectiveness of an anti-stigma intervention among primary care providers. Both staff and clients will be asked to complete survey data in order to measure the effectiveness. This is a randomized control trial in that three health centres will receive the intervention and three will not. Results will determine if this intervention reduces stigma among staff toward people with a mental health problem and/or substance use problem.

DETAILED DESCRIPTION:
The Office of Transformative Global Health at the Centre for Addiction and Mental Health (CAMH), with funding provided by the Canadian Institutes of Health Research (CIHR), has developed and will be implementing a three year anti-stigma study. This project is a randomized control study which compares the effectiveness of an anti-stigma intervention in three Toronto community health centres. Six centres were selected and randomized so that three receive the intervention and the other three do not. The goal is to determine if the intervention impacts service providers' attitudes and behaviours towards people with mental health problems and addictions. Additionally, the study measures client's perceptions of stigma in order to see if they believe stigma has been reduced or eliminated. The interventions incorporate the following components: innovative contact-based training, raising awareness, recovery-based arts, and a thorough analysis of each centre's policies and procedures.

Innovative contact-based training utilizes an adult education model and focuses on the results of a preliminary situational assessment conducted at each site. Emphasis is placed on concurrent disorders, cultural issues, and inter-professional collaboration. Four three-hour workshops were held at each intervention CHC throughout the project period and included a needs-based curriculum, contact-based education to reduce prejudice and social intolerance, and culturally competent care for vulnerable populations. Raising awareness includes various forms of media such as posters to increase awareness about stigma.

Recovery-based arts was geared towards a local team of leaders who selected one art form for their CHC and were taught by an art expert. Approximately ten service users with a mental health and/or substance abuse problem were invited to participate along with three staff members. After 10 bi-weekly art workshops, staff and clients will showcase their work at each CHC. Finally, an analysis of policies and procedures have been conducted by research staff. This determines what already exists and using an anti-stigma/pro-recovery approach to identify strengths and areas for improvement. Program and policies were studied to identify unintended positive and negative impacts using a modified version of the Health Equity Assessment Tool. Features of the Quality Rights Tool Kit were also used. Recommendations from this process will be developed and shared with each CHC.

ELIGIBILITY:
Inclusion Criteria:

* Staff - all staff, no matter their position, is asked to participate.
* Clients - individuals reporting current or past mental illness and/or substance use problems (MHSUD) AND have received services or participate in any programming at the CHC

Exclusion Criteria:

* Staff - no exclusion criteria
* Clients - Clients under the age of 18 years, clients who do not have a MHSUD, or clients that are not safely able to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2014-05; Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Opening Minds Scale for Health Care Providers (OMS-HC) | 2 years
  The OMS-HC is a 20-item Canadian scale that was developed specifically to measure stigma among healthcare providers toward individuals with mental illness.This scale has good internal consistency (Cronbach's alpha = 0.82), satisfactory test-retest reliability, intra-class correlation (0.66; 95% CI: 0.54-0.75)59 and sensitivity to change.
Mental Illness: Clinicians Attitudes Scale (MICA) | 2 years
  MICA is a 16-item scale that was also designed to measure attitudes among healthcare workers toward individuals with mental illness.The MICA scale has good internal consistency (Cronbach's alpha = 0.79), with a test-retest reliability (concordance) of 0.80 (95% CI: 0.68-0.91).
Modified Borgadus Social Distance Scale | 2 years
  The Modified Borgadus Social Distance Scale is based on the Borgadus Social Distance Scale.Our study will use a modified six-item version of this scale, focusing specifically on persons with one key mental illness (schizophrenia) and one key addiction (heroin dependence).

CONTACTS AND LOCATIONS:
Overall Officials: Akwatu A Khenti, MA, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khenti A, Mann R, Sapag JC, Bobbili SJ, Lentinello EK, Maas MV, Agic B, Hamilton H, Stuart H, Patten S, Sanches M, Corrigan P. Protocol: a cluster randomised control trial study exploring stigmatisation and recovery-based perspectives regarding mental illness and substance use problems among primary healthcare providers across Toronto, Ontario. BMJ Open. 2017 Nov 20;7(11):e017044. doi: 10.1136/bmjopen-2017-017044. PMID 29162572
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital, fully affiliated with the University of Toronto, and a PAHO/WHO Collaborating Centre — http://www.camh.net/research